CLINICAL TRIAL: NCT00366444
Title: Multicenter Study to Evaluate the Analgesic Efficacy of XP21L in Subjects With Pain Following Bunionectomy Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xanodyne Pharmaceuticals (Industry)
Responsible Party: Gary Shangold, MD / Chief Medical Officer, Xanodyne Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XP21L-301
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Results first posted 2011-04-13 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Pain, Postoperative
Keywords: Bunionectomy; Bunion surgery; Post-operative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Diclofenac

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: diclofenac potassium (XP21L)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: diclofenac potassium (XP21L) — 25 mg every 6 hours
  Other Names: Zipsor Liquid Filled Capsule; XP21L
  Arms: 1
Drug: Placebo — Placebo every 6 hours
  Arms: 2

SUMMARY:
A multicenter study to evaluate the analgesic efficacy of XP21L in subjects with pain following bunionectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Have undergone bunionectomy surgery
* Have achieved adequate post-surgical pain

Exclusion Criteria:

* Confounding medical conditions which preclude study participation
* Participated in a study of another investigational drug or device within 30 days prior to randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2006-08; Primary Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Investigative Site, Anaheim, California
  - Investigative Site, Orange, California
  - Investigative Site, Owings Mills, Maryland
  - Investigative Site, Pasadena, Maryland
  - Investigative Site, Altoona, Pennsylvania
  - Investigative Site, Salt Lake City, Utah

REFERENCES:
- [Result] Riff DS, Duckor S, Gottlieb I, Diamond E, Soulier S, Raymond G, Boesing SE. Diclofenac potassium liquid-filled soft gelatin capsules in the management of patients with postbunionectomy pain: a Phase III, multicenter, randomized, double-blind, placebo-controlled study conducted over 5 days. Clin Ther. 2009 Oct;31(10):2072-85. doi: 10.1016/j.clinthera.2009.09.011. PMID 19922878
- [Derived] Daniels SE, Riff D, Diamond E, Clark F, Boesing SE. An assessment of the efficacy and safety of diclofenac potassium liquid-filled capsules in patients with various levels of baseline pain intensity. Curr Med Res Opin. 2012 Jun;28(6):953-61. doi: 10.1185/03007995.2012.694363. Epub 2012 Jun 11. PMID 22587481
- See also: Related Info — http://www.xanodyne.com/pdf/results_disclosure.pdf.
- See also: Related Info — http://www.zipsor.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Zipsor (Diclofenac Potassium) Liquid Filled Capsule: 25 mg capsule, every 6 hours
- Placebo: Oral placebo capsule, every 6 hours
Period: Overall Study
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Started | 102 | 99
Completed | 101 | 97
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo | Total
Number analyzed (Participants) | 102 | 99 | 201
Age Continuous [Mean (Standard Deviation); unit: years] | 45 (11) | 45 (12) | 45 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 86 | 174
  Male | 14 | 13 | 27
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 61 | 56 | 117
  Black | 23 | 19 | 42
  Asian | 4 | 5 | 9
  Hispanic | 13 | 16 | 29
  Other | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 102 | 99 | 201
Baseline pain score [Mean (Standard Deviation); unit: units on a scale] — Pain intensity scores were measured using an 11-point numerical pain rating scale (NPRS) with 0=no pain to 10=worst possible pain
  units on a scale | 6.9 (1.7) | 7.3 (1.9) | 7.1 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Average Numeric Pain Rating Score (NPRS) Over 48 Hours After Bunionectomy
Description: Pain intensity scores were measured using an 11-point numerical pain rating scale (NPRS) with 0=no pain to 10=worst possible pain
Time Frame: Over 48 hours after bunionectomy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 102 | 99
units on a scale | 2.5 (2.0) | 5.6 (2.0)

2. Secondary Outcome: Number of Patients With Perceptible Pain Relief on Day 1
Description: Times to onset of Perceptible and Meaningful Relief were determined using the double-stopwatch method.
Time Frame: 8 hours post single dose
Measure: Number; unit: participants
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 102 | 99
participants | 84 | 69

3. Secondary Outcome: Median Time to Onset of Pain Relief in Patients With Perceptible Pain Relief on Day 1
Time Frame: 8 hours post single dose
Population: Number of participants analyzed includes only the number of participants with perceptible pain relief on Day 1 (see previous Outcome Measure #2)
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 84 | 69
minutes | 26.0 [18.6 to 31.3] | 22.2 [16.6 to 35.8]

4. Secondary Outcome: Number of Patients With Meaningful Pain Relief on Day 1
Description: Times to onset of Perceptible and Meaningful Relief were determined using the double-stopwatch method.
Time Frame: 8 hours post single dose
Measure: Number; unit: participants
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 102 | 99
participants | 58 | 35

5. Secondary Outcome: Median Time to Onset of Pain Relief in Patients With Meaningful Pain Relief on Day 1
Time Frame: 8 hours post single dose
Population: Number of participants analyzed includes only the number of participants with meaningful pain relief on Day 1 (see previous outcome measure, #4).
  Number of patients in the placebo group is intentionally blank as the data was not calculable since less than 50% of the patients reported meaningful relief (ie, median cannot be calculated).
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 58 | 0
minutes | 70.2 [61.2 to 92.0] |

6. Secondary Outcome: Total Pain Relief (TOTPAR) Scores 8 Hours Post Initial Dose of Study Drug
Description: Pain relief was rated using a 5-point categorial scale (0=none, 1=a little, 2=some, 3=a lot, and 4=complete) at time of dose (time=0) and over 15 time points afterwards (10, 15, 20, 30, 45, and 60 minutes and at 1.5, 2, 2.5, 3, 4, 5, 6, 7, and 8 hours after the initial dose on Day 1 or until time of re-medication). A score of 0 across all time points would be the lowest (worst) and a score of 60 (4 X 15 time points) would be the highest (best) possible score.
Time Frame: 8 hours post single dose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 102 | 99
units on a scale | 8.2 (9.3) | 2.6 (3.9)

7. Secondary Outcome: Number of Patients With at Least 30% Reduction in Pain Intensity After First Dose of Study Drug
Time Frame: 8 hours post single dose
Measure: Number; unit: participants
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 102 | 99
participants | 62 | 40

8. Secondary Outcome: Time to Onset of at Least 30% Reduction in Pain Intensity After First Dose of Study Drug
Time Frame: 8 hours post single dose
Population: Number of participants analyzed includes only the number of participants with at least a 30% reduction in pain intensity after the 1st dose (see previous outcome measure, #7).
  Number of placebo patients is intentionally blank as the data (eg., upper CI) was not calculable.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 62 | 0
minutes | 60 [45 to 90] |

9. Secondary Outcome: Number of Patients Who Required Rescue Medication on Day 1
Time Frame: Day 1
Measure: Number; unit: participants
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 102 | 99
participants | 40 | 87

10. Secondary Outcome: Number of Patients Who Required Rescue Medication on Day 2
Time Frame: Day 2
Measure: Number; unit: participants
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 102 | 99
participants | 22 | 64

11. Secondary Outcome: Number of Patients Who Required Rescue Medication on Day 3
Description: Day 3 data reflect the use of rescue medication only up to the time of discharge
Time Frame: Day 3
Measure: Number; unit: participants
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 102 | 99
participants | 5 | 29

ADVERSE EVENTS:
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Serious Adverse Events (participants affected / at risk) | 0/102 | 1/99
Other Adverse Events (participants affected / at risk) | 21/102 | 44/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zipsor (Diclofenac Potassium) Liquid Filled Capsule (N=102) | Placebo (N=99)
Superficial cellulitis of the left knee (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zipsor (Diclofenac Potassium) Liquid Filled Capsule (N=102) | Placebo (N=99)
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 4 | 2
Diarrhea (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 8 | 18
Vomiting (Gastrointestinal disorders) | 4 | 9
Body Temperature Increased (Investigations) | 0 | 3
Headache (Nervous system disorders) | 6 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3
Pyrexia (General disorders) | 0 | 8
Dizziness (Nervous system disorders) | 1 | 4
Anxiety (Psychiatric disorders) | 0 | 3
Hypertension (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other